CLINICAL TRIAL: NCT07062432
Title: Evaluating the Efficacy of a Continuous Comprehensive Nursing System on Postoperative Hemoglobin Levels and Quality of Life in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Continuous Comprehensive Nursing for Post-CABG Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Beibei Xing, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-HBLS-ky038
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: Continuous comprehensive nursing system; Coronary artery bypass surgery; Hemoglobin levels; Quality of life; Nursing Efficacy
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Comprehensive Nursing (CCN) System (Experimental): Participants received a continuous comprehensive care plan delivered by specifically trained cardiac nurses. This plan included:
  * Preoperative Phase: Comprehensive education about the surgery, risks, and expected outcomes, along with psychological support.
  * Intraoperative Phase: Standard intraoperative nursing care including close monitoring.
  * Postoperative Inpatient Phase: In addition to routine care, this phase focused on pain management, wound care, and individualized rehabilitation guidance.
  * Post-Discharge Continuous Phase (3 months): This phase included regular follow-up (monthly phone calls, one outpatient visit at 6 weeks), ongoing psychological support, continuous education (medication adherence, diet, activity), structured home-based rehabilitation training, and periodic evaluation of quality of life.
  Interventions: Behavioral: Continuous Comprehensive Nursing System
- Routine Care (Active Comparator): Participants received standard institutional postoperative care for CABG, which primarily focused on the inpatient period. Key elements included:
  * Monitoring of vital signs, consciousness, and peripheral circulation.
  * Management of respiratory tract patency and urinary catheters.
  * Hourly monitoring of drainage tubes initially.
  * Wound care and monitoring for bleeding.
  * Body temperature monitoring and oral care.
  * Guidance on progressing from liquid diets.
  * Standard discharge instructions without structured post-discharge follow-up.
  Interventions: Other: Routine Postoperative Care

INTERVENTIONS:
Behavioral: Continuous Comprehensive Nursing System — A multi-faceted nursing plan delivered by trained cardiac nurses, extending from the preoperative phase to 3 months post-discharge. In addition to routine inpatient care, the intervention included: preoperative education and psychological support; postoperative individualized rehabilitation guidance; and a continuous post-discharge program. The post-discharge phase involved structured follow-up (monthly phone calls, one 6-week outpatient visit), ongoing psychological support, reinforcement of education on medication adherence, diet, and activity progression, and guidance on a structured home-based exercise program.
  Arms: Continuous Comprehensive Nursing (CCN) System
Other: Routine Postoperative Care — Standard institutional postoperative care for patients after Coronary Artery Bypass Graft (CABG) surgery. This care was primarily focused on the inpatient period and included monitoring of vital signs, wound and drainage tube management, respiratory and circulatory support, and progressive diet guidance. The care concluded with standard discharge instructions and did not include the structured, continuous, or extended follow-up provided to the intervention group.
  Arms: Routine Care

SUMMARY:
This study evaluates the effectiveness of a continuous comprehensive nursing (CCN) system compared to routine care for patients after coronary artery bypass graft (CABG) surgery. The primary goal is to determine if the CCN system improves postoperative hemoglobin levels. The study also investigates the effects on quality of life, mental health (anxiety and depression), red blood cell indices, immune markers, and patient satisfaction.

DETAILED DESCRIPTION:
Coronary artery bypass surgery (CABG) is a major procedure, and the postoperative recovery process is complex, often impacting patients' hemoglobin levels and quality of life. Standard nursing care is often limited to the inpatient period. A continuous comprehensive nursing (CCN) system is a holistic, patient-centered model that extends care beyond hospital discharge. This model includes preoperative education, continuous monitoring, personalized care plans, psychological support, rehabilitation guidance, and structured follow-up. While the benefits of comprehensive nursing are recognized, its specific impact on hemoglobin recovery and quality of life after CABG has not been extensively studied. This randomized controlled trial was designed to compare the outcomes of patients receiving a CCN plan with those receiving routine postoperative care to provide evidence for optimizing post-CABG nursing strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Confirmed diagnosis of coronary heart disease and evidence of coronary artery illness requiring CABG.
* Ability to understand the purpose and procedures of the study.
* Willingness to sign the informed consent form.

Exclusion Criteria:

* Presence of serious complications such as unstable myocardial ischemia or significant arrhythmia.
* Severe lung diseases (e.g., chronic obstructive pulmonary disease GOLD stage III/IV).
* Severe kidney diseases (e.g., chronic kidney disease Stage 4/5).
* Significantly impaired left ventricular ejection fraction (EF < 30%).
* Concurrent participation in other clinical trials or receiving other interventions.
* Presence of severe mental illnesses or cognitive impairments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin (Hb) Levels from Baseline to Day 7 Post-Surgery | Baseline (preoperatively) and Day 7 post-surgery.
  The change in hemoglobin concentration (g/L) was measured from the preoperative baseline value to the value at 7 days after the surgery. Venous blood samples were analyzed using an automatic biochemical analyzer.

SECONDARY OUTCOMES:
Change in Hemoglobin (Hb) Levels at Other Time Points | Baseline, 12 hours, 72 hours, and 14 days post-surgery.
  Hemoglobin concentration (g/L) measured at multiple time points to assess the recovery trajectory.
Red Blood Cell Indices | Day 7 post-surgery.
  Measurement of Mean Corpuscular Volume (MCV, in fL), Red Blood Cell Distribution Width (RDW, in %), and Hematocrit (HCT, in %).
Levels of Immune-Related Inflammatory Markers | Day 7 post-surgery.
  Levels of Interleukin-2 (IL-2, in pg/mL) and Interleukin-6 (IL-6, in pg/mL) in peripheral blood, quantified using an ELISA kit.
Quality of Life (QoL) | Day 14 post-surgery.
  Assessed using the World Health Organization Quality of Life BREF (WHOQOL-BREF) scale. This scale evaluates four domains: physical health, psychological health, social relationships, and environment. Higher scores indicate better quality of life.
Depressive Symptoms | Day 14 post-surgery.
  Assessed using the Center for Epidemiologic Studies Depression Scale (CES-D). The scale ranges from 0 to 60, with higher scores indicating more severe depressive symptoms.
Anxiety Symptoms | Day 14 post-surgery.
  Assessed using the Self-Rating Anxiety Scale (SAS). The scale ranges from 20 to 80, with higher scores reflecting more severe anxiety symptoms.
Patient Satisfaction | Up to 14 days post-surgery (at time of hospital discharge).
  Assessed using a study-specific satisfaction questionnaire. Responses were categorized as "very satisfied," "satisfied," "average," or "dissatisfied" based on a scoring system from 1-100.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China